CLINICAL TRIAL: NCT05766267
Title: Phase 2C Clinical Trial of Novel, Short-course Regimens for the Treatment of Pulmonary Tuberculosis: CRUSH-TB (Combination Regimens for Shortening TB Treatment)
Brief Title: Short-course Regimens for the Treatment of Pulmonary Tuberculosis
Acronym: CRUSH-TB
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Tuberculosis Trials Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7406
Record Dates: First submitted 2022-10-05; First posted 2023-03-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis Infection
MeSH Terms: conditions — Tuberculosis, Pulmonary; Latent Tuberculosis | interventions — Rifabutin; OPC-67683; bedaquiline; Moxifloxacin; Pyrazinamide; Isoniazid; Rifampin; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2BMZRb/2 BMRb (Experimental): Eight weeks of daily treatment with bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), plus rifabutin (Rb), followed by nine weeks of daily treatment with bedaquiline (B or BDQ), moxifloxacin (M) and Rifabutin (Rb)
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered once daily.
  Study drug doses: Bedaquiline (B): 200 mg once daily x 56 days, then 100 mg daily; Moxifloxacin (M): 400 mg once daily; Pyrazinamide (Z) 1500 mg (weight <75kg) or 2000mg(> 75kg) once daily x 56 days; Rifabutin (Rb): 300 mg once daily
  Interventions: Drug: Rifabutin; Drug: Bedaquiline; Drug: Moxifloxacin; Drug: Pyrazinamide
- 2 BMZD/2 BMD (Experimental): Eight weeks of daily treatment with bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), plus delamanid (D or DLM) followed by nine weeks of daily treatment with bedaquiline (B or BDQ), moxifloxacin (M) and delamanid (D or DLM)
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered once daily.
  Study drug doses: Bedaquiline (B): 200 mg once daily x 56 days, then 100 mg daily; Moxifloxacin (M): 400 mg once daily; Pyrazinamide (Z) 1500 mg (weight <75kg) or 2000mg(> 75kg) once daily x 56 days; Delamanid (D):300 mg once daily
  Interventions: Drug: Delamanid; Drug: Bedaquiline; Drug: Moxifloxacin; Drug: Pyrazinamide
- 2RHZE/4RH (Active Comparator): Eight weeks of daily treatment with rifampin, isoniazid, pyrazinamide, and ethambutol, followed by eighteen weeks of daily treatment with rifampin and isoniazid
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered once daily
  study drug doses: Rifampin (R), 600 mg daily; Isoniazid (H), 300 mg daily; Pyrazinamide (Z) 1500 mg (weight <75kg) or 2000mg(> 75kg) once daily ; Ethambutol, 15 mg/kg once daily rounded up to nearest 400 mg dose
  Interventions: Drug: Pyrazinamide; Drug: Isoniazid; Drug: Rifampin; Drug: Ethambutol

INTERVENTIONS:
Drug: Rifabutin — Rifabutin (Rb) is added to the bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), (BMZ) regimen for first 8 weeks and continued for next 9 weeks with bedaquiline (B or BDQ) and moxifloxacin (M)
  Arms: 2BMZRb/2 BMRb
Drug: Delamanid — Delamanid (D or DLM) is added to the bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), (BMZ) regimen for first 8 weeks and continued for next 9 weeks with bedaquiline (B or BDQ) and moxifloxacin (M)
  Other Names: Deltyba
  Arms: 2 BMZD/2 BMD
Drug: Bedaquiline — Bedaquiline is part of interventional arms with bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z)-- (BMZ).
  Other Names: Sirturo
  Arms: 2 BMZD/2 BMD; 2BMZRb/2 BMRb
Drug: Moxifloxacin — Moxifloxacin is part of interventional arms with bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z)-- (BMZ).
  Arms: 2 BMZD/2 BMD; 2BMZRb/2 BMRb
Drug: Pyrazinamide — Pyrazinamide is part of interventional arms with bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z)-- (BMZ). Pyrazinamide is part of control regimen (HRZE).
Drug: Isoniazid — Isoniazid is part of control regimen (HRZE).
  Arms: 2RHZE/4RH
Drug: Rifampin — Rifampin is part of control regimen (HRZE).
  Arms: 2RHZE/4RH
Drug: Ethambutol — Ethambutol is part of control regimen (HRZE).
  Arms: 2RHZE/4RH

SUMMARY:
The purpose of this study is to determine whether one or two 17-week regimens of tuberculosis treatment bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z)-- (BMZ) plus either Rifabutin (Rb) or Delamanid (D or DLM) are as effective as a standard six-month regimen for treatment of pulmonary tuberculosis (TB). All three regimens are administered daily, seven days each week.

The first 17-week regimen is 2 months of bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), (BMZ) plus rifabutin (Rb) (BMZRB) followed by 2 months of bedaquiline (B or BDQ), moxifloxacin (M) and Rifabutin (Rb) (2 BMZRb/2 BMRb, Arm 1)

The Second 17-week regimen is 2 months of bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), (BMZ) plus delamanid (D or DLM); (BMZD) followed by 2 months of bedaquiline (B or BDQ), moxifloxacin (M) and delamanid (D or DLM) (2 BMZD/2 BMD, Arm 2)

The standard 26-week treatment control regimen which is two months of isoniazid, rifampin, ethambutol, and pyrazinamide (2HRZE) followed by four months of isoniazid and rifampin (4HR); (2HRZE/4HR, Arm 3)

Target enrollment is 288 male and female participants (96/arm). participants. Participants will be followed until 78 weeks post-randomization, or until the last enrolled participant completes 52 weeks post-randomization, whichever comes first.

DETAILED DESCRIPTION:
Phase 2C Clinical Trial of Novel, Short-course Regimens for the Treatment of Pulmonary Tuberculosis: CRUSH-TB (Combination Regimens for Shortening TB Treatment)

Hypotheses:

1. The time to sputum culture negative in liquid media will be shorter in the 17-week regimen of 2 months of bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), (BMZ) plus rifabutin (Rb) followed by 2 months of bedaquiline (B or BDQ), moxifloxacin (M) and Rifabutin (Rb) (2BMZRb/2 BMRb, Arm 1) than in the control arm.
2. The time to sputum culture negative in liquid media will be shorter in the 17-week regimen of 2 months of bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z); (BMZ) plus delamanid (D or DLM) followed by 2 months of bedaquiline (B or BDQ), moxifloxacin (M) and delamanid (D or DLM) (2 BMZD/2 BMD, Arm 2) than in the control arm.

Phase: 3 Design: Open label, randomized clinical trial, initially in three treatment groups, with adaptive design allowing for introduction of novel regimens once they are clinically ready for testing Population: newly diagnosed with sputum smear positive or GeneXpert positive pulmonary tuberculosis, aged 12 years or older, with normal QTcF (QTc interval, Fridericia calculation) on screening ECG.

Number of Sites: 13 National and International sites, primarily sites of the Tuberculosis Trials Consortium Group. Study Duration: Duration per participant is approximately 78 weeks Description of Agent or Intervention: After written informed consent, participants will be randomized 1:1:1 to receive BMZRb, BMZD, or HRZE (Control treatment) as below

Arm 1(investigational regimen): 2 BMZRb/2 BMRb

* Eight weeks of daily treatment with bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), plus rifabutin (Rb), followed by
* Nine weeks of daily treatment with bedaquiline (B or BDQ), moxifloxacin (M) and Rifabutin (Rb)

Arm 2 (investigational regimen): 2 BMZD/2 BMD

* Eight weeks of daily treatment with bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), plus delamanid (D or DLM) followed by
* Nine weeks of daily treatment with bedaquiline (B or BDQ), moxifloxacin (M) and delamanid (D or DLM)

Arm 3 (Control regimen): 2 RHZE/4 RH

* Eight weeks of daily treatment with rifampin (R), isoniazid (H), pyrazinamide (Z), and ethambutol (E), (RHZE) followed by
* Eighteen weeks of daily treatment with rifampin and isoniazid (RH)

Objectives

Primary Objectives:

1. To compare the efficacy of 17-week regimen 8 weeks of bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), (BMZ) plus rifabutin (Rb) followed by 9 weeks of bedaquiline (B or BDQ), moxifloxacin (M) and rifabutin (Rb) (2 BMZRb/2 BMRb) experimental regimen to the efficacy of standard treatment, using the intermediate endpoint of time to culture negative in liquid media.
2. To compare the efficacy of 17-week regimen 8 weeks of bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z), (BMZ) plus delamanid (D or DLM) followed by 9 weeks of bedaquiline (B or BDQ), moxifloxacin (M) and delamanid (D or DLM) (2 BMZD/2 BMD) experimental regimen to the efficacy of standard treatment, using the intermediate endpoint of time to culture negative in liquid media.

Secondary Objectives:

1. To compare the proportion of participants with a grade 3 or higher adverse event in each experimental arm with the control arm
2. To describe the proportion of participants experiencing lack of sustained cure during treatment or follow-up to 52 weeks in each experimental arm as compared to control and make predictions as to how these regimens would perform in future phase III trials.
3. To compare the efficacy of each experimental regimen to the efficacy of standard treatment, using the intermediate endpoint of time to culture negative in solid media
4. To compare the proportion of participants in each arm who convert liquid and solid sputum cultures to negative by (a) 8 weeks of treatment and (b) 12 weeks of treatment
5. To describe the rate of all-cause study drug discontinuation in each arm
6. To compare time to sputum culture positivity curves through 17 weeks in the Mycobacterial Growth Indicator Tube (Bactec MGIT960) across arms
7. To describe the proportion of participants experiencing lack of sustained cure during treatment or follow-up up to 78 weeks in each experimental arm as compared to control and make predictions as to how these regimens would perform in future phase III trials.
8. To describe the population PK of bedaquiline and its M2 metabolite, with or without rifabutin co-administration (PK#1)
9. To conduct pharmacokinetic/pharmacodynamics study of the test drugs to determine relationships between pharmacokinetic parameters (AUC, Cmax) and outcome measures (time to culture negativity or rate of change in TTP) using non-linear mixed effects models, adjusting for key covariates that may affect outcomes (e.g. companion drugs, HIV status, cavitary disease) (PK#2)

Primary Endpoints:

1. Time to sputum culture negative in liquid media

Secondary Endpoints:

1. Proportion of participants with a Grade 3 or higher adverse event during 26 weeks from randomization
2. Lack of sustained cure during treatment or follow-up to 52 weeks
3. Time to sputum culture negative in solid media
4. Proportion of participants with sputum culture negative by 8 weeks and by 12 weeks (solid and liquid media).
5. All-cause study drug discontinuation
6. The rate of change in time to sputum culture positivity (TTP) through 17 weeks in the Mycobacterial Growth Indicator Tube (Bactec MGIT960)
7. Lack of sustained cure during treatment or follow-up to 78 weeks
8. Population pharmacokinetics (PK) of bedaquiline, with or without rifabutin Pharmacokinetic/pharmacodynamic (PK/PD) relationship between test drug PK parameters and microbiologic outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary tuberculosis with or without suspected or proven concomitant extrapulmonary tuberculosis outside the central nervous system or bones
2. Acid-fast bacilli (AFB) seen in an expectorated sputum specimen at least 1+ or positive GeneXpert (or GeneXpert Ultra) for M. tuberculosis, with semiquantitative results of "medium" or "high".
3. Age ≥12 years
4. Documentation of negative HIV status within the past 3 months prior to enrollment or documentation confirming HIV infection.
5. For participants with HIV:

   1. current use of dolutegravir-based ART (Anti Retroviral Therapy), or ability and willingness to start or transition to a dolutegravir-based antiretroviral therapy regimen
   2. CD4 T cell count greater than or equal to 100 cells/mm3 based on testing performed at or within 30 days prior to study enrollment
6. Written informed consent/assent
7. Karnofsky score of at least 60 ("requiring some help, can take care of most personal requirements")
8. A verifiable address or residence location that is readily accessible for visiting, and willingness to inform the study team of any change of address during the treatment and follow-up period.
9. For all women who have not undergone a surgical sterilization procedure or who do not meet the study definition of post-menopausal, a negative pregnancy test at or within seven (7) days prior to screening
10. For all individuals of child-bearing potential who are not surgically sterilized, agreement to practice a reliable method of contraception (barrier method or non-hormonal intrauterine device) or abstain from sexual activity that could lead to pregnancy while receiving study drug treatment and for 30 days after stopping study treatment

Exclusion Criteria:

1. Pregnant or breast-feeding
2. More than 5 days of tuberculosis treatment in the previous 6 months
3. Previous treatment with any drug or combination of drugs known to have activity against M. tuberculosis (e.g., isoniazid, rifamycins, pyrazinamide, ethambutol, fluoroquinolones, etc.) for more than five days in the thirty days prior to enrollment
4. Unable to take oral medications
5. Hypersensitivity or previous intolerance to any of the study drugs
6. Current or planned use of medications that have unacceptable drug-drug interactions with any of the study drugs during study treatment
7. Suspected or proven central nervous system tuberculosis
8. Suspected or proven bone tuberculosis
9. Screening ECG with QTcF >450 for men or >470 for women (Note: in case of hypokalemia or hypomagnesemia, ECG can be repeated following electrolyte supplementation)
10. Clinically significant ECG abnormality in the opinion of the site investigator, including but not limited to second or third degree atrioventricular (AV) block, prolongation of the QRS complex over 120 ms (in both male and female participants), or clinically important arrhythmia
11. Current clinically relevant cardiovascular disorder in the opinion of the site investigator, including but not limited to heart failure, coronary heart disease, arrhythmia, or tachyarrhythmia
12. Known family history of Long QT Syndrome in a first-degree relative (i.e., parent, offspring, or sibling)
13. History of aortic aneurysm or dissection
14. Hepatic cirrhosis or other serious liver disease
15. Other medical conditions, that, in the investigator's judgment, make study participation not in the individual's best interest.
16. Laboratory parameters done at or within 14 days prior to screening:

    1. Serum or plasma alanine aminotransferase greater than 3 times the upper limit of normal
    2. Serum or plasma total bilirubin greater than 2.5 times the upper limit of normal
    3. Serum creatinine > 2 times the upper limit of normal
    4. Platelet count < 75,000 cells/mm3
    5. Absolute neutrophil count <1,000 cells/mm3
    6. Serum or plasma potassium <3.5 meq/L (note: potassium may be repleted and test repeated)
17. Weight less than 40.0 kg
18. Known or suspected resistance to isoniazid or rifamycins (by phenotypic or molecular test)
19. Previously enrolled in this study or currently enrolled in another therapeutic clinical trial that, in the investigator's judgment, would compromise study integrity or participant safety
20. Current or planned incarceration or other involuntary detention.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to sputum culture negative in liquid media after study treatment among participants in Experimental Regimens (2 BZMRb/ 2 BMRb, Arm 1) and (2 BMZD/ 2 BMD, Arm 2) compared to Control (2HRZE/4HR, Arm 3) in modified intention-to-treat group (ITT) | 17 weeks
  The purpose of this study is to determine whether one or two 17-week regimens of tuberculosis treatment bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z)-- (BMZ) plus either Rifabutin (Rb) or Delamanid (D or DLM) are as effective as a standard six-month regimen for treatment of pulmonary tuberculosis (TB). All three regimens are administered daily, seven days each week. The time to culture negative will be defined as the time from randomization to the date of the first of at least two consecutive negative sputum cultures, collected on different study visits, irrespective of any subsequent positive cultures that may occur. Modified intention-to-treat group includes all participants in the ITT population (all enrolled participants who receive a treatment assignment) except late exclusions

SECONDARY OUTCOMES:
The proportion of participants with a grade 3 or higher adverse event in Experimental Regimens (2 BZMRb/2 BMRb, Arm 1) and (2 BMZD/2 BMD, Arm 2) compared to Control Regimen (2HRZE/4HR, Arm 3) in the modified intention-to-treat group | up to 78 weeks
  To evaluate the safety of one or two 17-week regimens of tuberculosis treatment bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z)-- (BMZ) plus either Rifabutin (Rb) or Delamanid (D or DLM) are as effective as a standard six-month regimen for treatment of pulmonary tuberculosis (TB). All three regimens are administered daily, seven days each week. Safety Analysis includes all participants in the ITT population that receive at least one dose of study medication
The proportion of participants experiencing lack of sustained cure in each experimental regimens (2BZMRb/2BMRb, Arm 1) and (2BMZD/2BMD, Arm 2) compared to Control Regimen (2HRZE/4HR, Arm 3) | up to 52 weeks
  Sustained Culture Negativity is achieved when a participant's last two culture results collected on different study visits are negative (without an intervening positive result), the last of which is collected no earlier than 48 weeks after randomization (allowing for a 4 week window prior to the 52 week timepoint
The proportion of participants experiencing lack of sustained cure in each experimental regimens (2BZMRb/2BMRb, Arm 1) and (2BMZD/2BMD, Arm 2) compared to Control Regimen (2HRZE/4HR, Arm 3) | up to 78 weeks
  Sustained Culture Negativity is achieved when a participant's last two culture results regimens (2BZMRb/2BMRb, Arm 1) and (2BMZD/2BMD, Arm 2) compared to Control Regimen (2HRZE/4HR, Arm 3)collected on different study visits are negative (without an intervening positive result), the last of which is collected no earlier than 48 weeks after randomization (allowing for a 4 week window prior to the 52 week timepoint
Time to sputum culture negative in solid media after study treatment assignment among participants in Experimental Regimens (2BZMRb/2BMRb, Arm 1) and (2BMZD/2BMD, Arm 2) compared to Control Regimen (2HRZE/4HR, Arm 3) in modified intention-to-treat group | up to 78 weeks
  The purpose of this study is to determine whether one or two 17-week regimens of tuberculosis treatment bedaquiline (B or BDQ), moxifloxacin (M), pyrazinamide (Z)-- (BMZ) plus either Rifabutin (Rb) or Delamanid (D or DLM) are as effective as a standard six-month regimen for treatment of pulmonary tuberculosis (TB). All three regimens are administered daily, seven days each week. The time to culture negative will be defined as the time from randomization to the date of the first of at least two consecutive negative sputum cultures, collected on different study visits, irrespective of any subsequent positive cultures that may occur. Modified intention-to-treat group includes all participants in the ITT population (all enrolled participants who receive a treatment assignment) except late exclusions
Proportion of participants with sputum culture negative by 8 weeks and by 12 weeks (solid and liquid media) in all 3 regimens | 8 weeks and 12 weeks
  The time to culture negative will be defined as the time from randomization to the date of the first of at least two consecutive negative sputum cultures, collected on different study visits, irrespective of any subsequent positive cultures that may occur
All-cause study drug discontinuation among participants in experimental regimens compared to control regimen | up to 26 weeks
  Any discontinuation in study treatment by the participant
The rate of change in time to sputum culture positivity (TTP) through 17 weeks in the Mycobacterial Growth Indicator Tube (Bactec MGIT960) among participants in all three regimens | 17 weeks
  rate of change in time to sputum culture positivity (TTP) through 17 weeks in the Mycobacterial Growth Indicator Tube (Bactec MGIT960) will be measured and compared
Clearance of bedaquiline | 17 weeks
  Population PK parameter, Clearance of bedaquiline with or without rifabutin co-administration, will be measured for each experimental arm
Volume of Distribution of bedaquiline | 17 weeks
  Population PK parameter, Volume of Distribution of bedaquiline with or without rifabutin co-administration, will be measured for each experimental arm
Rate of absorption of bedaquiline | 17 weeks
  Population PK parameter: rate of absorption of bedaquiline with or without rifabutin co-administration, will be measured for each experimental arm

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dooley, MD, Study Chair — Johns Hopkins University; Daniel W Fitzgerald, MD, Study Chair — Weill Medical College of Cornell University; Ekaterina V Kurbatova, MD, PhD, MPH, Study Chair — Centers for Disease Control and Prevention; Wendy Carr, PhD, Study Chair — Centers for Disease Control and Prevention
Locations (8):
- TBTC Site 26 Seattle & King County TB Control Program, Seattle, Washington, United States
- Canada (2):
  - McGill University Health Centre, Montreal
  - Vancouver, British Columbia Centre for Disease Control, Vancouver
- Haiti (2):
  - TBTC Site 67 GHESKIO centers IMIS, Port-au-Prince, Ouest
  - TBTC Site 45 Les Centres Gheskio (INLR), Port-au-Prince, Ouest
- TBTC Site 09 University of Cape Town Lung Institute (Pty) Ltd, Mowbray, Cape Town, South Africa
- TBTC Site 30 Uganda-Case Western Reserve Research Collaboration, Kampala, Uganda
- TBTC Site 76 CAB-V. Can Tho Province, Vietnam - Thot Not District TB Unit, Can Tho, Can Tho City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data being collected in CDISC format
Supporting Information: Study Protocol, ICF
Time Frame: After the study completion and during results submission
Access Criteria: Upon request

REFERENCES:
- [Derived] Kurbatova EV, Dooley KE, Carr W, Stout JE, Nuermberger EL, Phillips PPJ, Scott NA, Upton CM, Ignatius E, Haas M, Walter ND, Traxler RM, Brown NE, Boyd R, Bryant KE, Dixon MG, Savic R, Eichberg C, Hesseling A, Bark C, Benator DA, Muzanyi G, Twycross NS, Fox GJ, Pierre S, Burzynski J, Fitzgerald DW; TBTC Study 38 CRUSH-TB Team. Phase 2C clinical trial of novel short-course regimens for the treatment of pulmonary tuberculosis: TBTC study 38/CRUSH-TB design. Contemp Clin Trials. 2025 Nov;158:108075. doi: 10.1016/j.cct.2025.108075. Epub 2025 Sep 5. PMID 40915316